CLINICAL TRIAL: NCT06604481
Title: Randomized Controlled Trial to Test the Efficacy of Online Ecoaching to Support Caregivers of Older Adults in Hong Kong: Enhancing Carers' Wellbeing and Resilience
Brief Title: An Online Ecoaching RCT Intervention for Carers: Enhancing Wellbeing and Resilience Through Self-Help Strategies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Vivian W.Q. Lou, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-0030-001-e
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Caregiver Burden; Self Efficacy; Quality of Life; Anxiety Depression; Resilience
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eCoaching Group I (Experimental): Online intervention based on Cognitive Behavioral Therapy, Dialectical Behavioral Therapy, lifestyle intervention, and effective communication skills. All content will be covered.
  Interventions: Behavioral: eCoaching for Caregivers of Older Adults
- eCoaching Group II (Experimental): Online intervention based on Cognitive Behavioral Therapy, Dialectical Behavioral Therapy, lifestyle intervention, and effective communication skills. Content will be covered specified to the carer's specific needs.
  Interventions: Behavioral: eCoaching (need specific) for Caregivers of Older Adults
- Control Group (Active Comparator): Online sessions focused on education about lifestyle and communication.
  Interventions: Behavioral: Control Intervention for Caregivers of Older Adults

INTERVENTIONS:
Behavioral: eCoaching for Caregivers of Older Adults — The experimental group receives an online intervention based on Cognitive Behavioral Therapy, Dialectical Behavioral Therapy, lifestyle intervention, and effective communication skills. This program is designed to operate individually on an e-platform. It consists of 6 weekly sessions, each lasting for less than 90 minutes. The content of the sessions focuses on teaching caregivers CBT techniques, lifestyle modifications to improve caregiving experiences, and effective communication strategies. In between each session, participants are assigned home practices to reinforce the skills learned further. All content will be included.
  Arms: eCoaching Group I
Behavioral: eCoaching (need specific) for Caregivers of Older Adults — The experimental group receives an online intervention based on Cognitive Behavioral Therapy, Dialectical Behavioral Therapy, lifestyle intervention, and effective communication skills as in eCoaching I. However, eCoaching II will include content specified to carer's specific need.
  Arms: eCoaching Group II
Behavioral: Control Intervention for Caregivers of Older Adults — The control group attends 6 weekly online sessions that primarily provide educational information about lifestyle factors and communication. These sessions aim to enhance the control group's knowledge and understanding of the factors that impact caregiving. Each session in the control group also lasts for 90 minutes. The focus of these activities will be on building practical caregiving skills and promoting overall well-being, rather than targeting any particular psychological or mental health-related factors directly.
  Arms: Control Group

SUMMARY:
The goal of this three-armed, double-blind randomized controlled trial (RCT) is to compare the effectiveness of an online self-help eCoaching intervention designed for caregivers. The main questions it aims to answer are:

What is the impact of the online self-help eCoaching intervention on the well-being, depressive symptoms, and self-efficacy of participants? Researchers will compare the results between the intervention groups and the control group to see if participants in the intervention groups have lower distress, burden and higher accuracy.

DETAILED DESCRIPTION:
Proposed Study:

The investigators propose a 6-week randomized controlled trial to compare the effectiveness of a novel online self-help intervention for caregivers of older adults in Hong Kong. The intervention is based on Cognitive Behavioral Therapy, lifestyle intervention, and effective communication skills.

Randomization:

The research team will perform individual randomization using statistical software R. Randomization will be using random permuted blocks via an online computer randomization system from an independent clinical trials unit. Participants will be randomized into two intervention groups or control group.

Outcomes:

The primary objective of this study is to evaluate the effectiveness of an online self-help eCoaching intervention that incorporates symptom management, stress management, and coping skills training in promoting healthy behavior change among caregivers. Additionally, this study aims to investigate the effectiveness of the online self-help eCoaching intervention in reducing carers' depressive symptoms and anxiety. Another key objective is to enhance carers' self-efficacy for stress management and resilience by equipping them with the necessary skills and strategies provided through the eCoaching intervention.

Recruitment and Inclusion Criteria:

A total of 232 caregivers from seven district-based caregiver support units will be recruited. The inclusion criteria are as follows: 1) Participants must be adults aged 18 or above with a family member aged 60 or above requiring caregiving, providing at least 6 hours of care per week; 2) They must self-identify as a family caregiver; 3) Participants must live in Hong Kong and 4) be able to communicate with the interventionist; 5) Participation must be voluntary; 6) Additionally, participants must report mild need in the Carer multidimensional Need Assessment tool. The exclusion criteria include: 1) having diagnosed Alzheimer's or other dementia; or 2) experiencing acute health conditions that hinder caregiving support or intervention participation.

Study Procedures:

This study will consist of a 6-week intervention, with a screening process to be conducted prior to the intervention implementation. Baseline and immediately after the intervention, as well as a 3-month follow-up assessment, will be performed for statistical comparison. The participation of caregivers in tests, surveys, and interviews will not affect the quality of care they receive. No drug usage or medical treatment is involved in this study, and there are no anticipated physical or medical risks to participants. Withdrawal from the study is voluntary at any time, and will not impact participants' ongoing medical care or legal rights.

The screening process involves carers completing a standardized screening form comprising items pertaining to demographics, self-efficacy, caregiving preparedness, and willingness to join, which they will either fill out independently or have facilitated by project staff upon enrolling for membership. Carers' needs are classified into four levels: low, mild, moderate, and high.

The Carer Multidimensional Need Assessment Tool was developed and validated by the research team of the Jockey Club Carer Space Project, which was led by Professor Vivian Lou, the Director of the Sau Po Centre on Ageing at the University of Hong Kong. The research centre followed a six-step approach, based on the scale development method proposed by Hinkin (1995), to establish the Carer Need Screening Tool. These steps encompassed: (1) a literature review, (2) the formation of an expert panel, (3) a Delphi study, (4) the confirmation of an item list, (5) an item validation study, and (6) the finalization of the scale. The research team developed a 22-item screening tool, and the screening tool involves 5 domains of risk including carers' mental ill health, caregiving capacity, lack of support, carers' health challenges, and high care demands.

Data Analysis:

A MANOVA will be conducted for the continuous variables and a chi-square test will be used for the categorical variables, to compare the differences between the primary and secondary outcomes of the three groups. The associations among different variables will be investigated using Pearson's correlation analysis. The interaction Group x Time treatment effects within and between the groups (eCoaching I, eCoaching II, Control) will be tested with a factorial ANOVA with repeated measures. Differential changes in each outcome across the 3 assessment time points (T0, T1, T2) between the three treatment groups will be compared. Recruitment rate, attrition rate, and missing data will also be examined and reported. All outcome measures will be analysed based on intention-to-treat principles. Exploratory analysis will assess whether the intervention effects are mediated by caregiver self-efficacy or knowledge gain. The data will be analysed using SPSS, version 28.0. All statistical tests will be two-sided with the level of significance set at .05.

Data Storage and Privacy:

Personal data will be securely stored by the principal investigator for 5 years after the publication of the first paper, followed by 10 years for anonymized data. All information will be used for research purposes only and stored on encrypted workstations and password-protected online cloud storage.

ELIGIBILITY:
Inclusion Criteria:

* being an adult aged 18 or above with a family member aged 60 or above requiring caregiving, providing at least 6 hours of care per week
* self-identifying as a family caregiver
* living in Hong Kong
* able to communicate with the interventionist
* voluntary participation
* reporting mild risk need in Carer Need Screening tool

Exclusion Criteria:

* having diagnosed Alzheimer's or other dementia
* experiencing acute health conditions that hinder caregiving support or intervention participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 3 months
  The PHQ-9 is a self-report instrument used to assess symptoms of depression.
Carers Multidimensional Need Assessment Tool | 3 months
  Carers Multidimensional Need Assessment Tool 22-item. The Carers Multidimensional Need Assessment Tool is a 22-item assessment that evaluates caregivers across 5 key domains of risk:Carers' mental ill health, Caregiving capacity, Lack of support, Carers' health challenges and High care demands.
Generalised Anxiety Disorder (GAD-7) | 3 months
  The GAD-7 is a 7-item screening tool used to assess the severity of generalized anxiety disorder.

SECONDARY OUTCOMES:
Cantonese short version of the Zarit Burden Interview (CZBI) | 3 months
  Reduced burden of caregivers
The World Health Organization Quality of Life (WHOQoL-BREF) | 3 months
  The WHOQOL-BREF is a 28-item instrument developed by the World Health Organization to assess an individual's quality of life across four domains: physical health, psychological health, social relationships, and environment.
Connor-Davidson Resilience Scale (CD-RISC-25) | 3 months
  The CD-RISC is a 25-item self-administered scale that assesses an individual's level of resilience.
Self-Care Self-Efficacy Scale (SCSES-10) | 3 months
  The SCSES-10 is a measurement tool used to assess an individual's self-efficacy self-care self-efficacy for chronic illness and has been tested in the Hong Kong population.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Lou, PhD, Principal Investigator — Sau Po Center on Ageing, HKU
Locations (1):
- Sau Po Center on Ageing HKU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be published and submitted to academic journals to share with other researchers.
Supporting Information: Study Protocol
Time Frame: Between 2024 and 2026, the data will become available.
Access Criteria: Upon request from the academic journals.